CLINICAL TRIAL: NCT01417091
Title: A Randomized, Open Label Intra-patient Dose Escalation Study With an Untreated Reference Group to Evaluate Safety and Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Infusions of BPS804 in Adults With Moderate Osteogenesis Imperfecta
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of BPS804 in Osteogenesis Imperfecta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBPS804A2201; 2011-001465-41 (EudraCT Number)
Record Dates: First submitted 2011-08-04; First posted 2011-08-16 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Osteogenesis Imperfecta
Keywords: Brittle bone disease; inherited; connective tissue disorder; fracture
MeSH Terms: conditions — Osteogenesis Imperfecta; Connective Tissue Diseases; Fractures, Bone | interventions — setrusumab

ARMS (2):
- Treatment group (Experimental)
  Interventions: Drug: BPS804
- Untreated reference group (No Intervention)

INTERVENTIONS:
Drug: BPS804
  Arms: Treatment group

SUMMARY:
This is a randomized, open label intra-patient dose escalation study to evaluate safety and tolerability, pharmacokinetics, and pharmacodynamics of BPS804 in adults with osteogenesis imperfecta (OI).

Pharmacodynamic effect will be determined by serological biomarkers and radiologic assessments. In addition, tolerability and pharmacokinetics (PK) will be evaluated.

DETAILED DESCRIPTION:
This study was previously posted by Mereo BioPharma and was transferred to Ultragenyx in February 2021.

ELIGIBILITY:
Inclusion Criteria:

* Osteogenesis imperfecta
* Two or more previous fractures
* Bone mineral density Z-score of ≤ -1.0 and > -4.0

Exclusion Criteria:

* Open epiphyses
* Fracture within last 2 weeks
* Treatment with bisphosphonates/teriparatide (last 6 months)
* Surgery within last year

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (composite outcome: standard laboratory, (serious) adverse events) | Day 1 through 141
  The assessment of safety will be based on primarily on the frequency of adverse events, laboratory abnormalities, and serious adverse events suspected by the investigators to be related to study treatments. The AE collection period extends from the time of first study drug administration drug until study completion. The intensity of each AE will be characterized and classified into 1 of the 3 generic categories (mild, moderate, or severe). The number and percentage of patients with adverse events will be tabulated by treatment group, body system and preferred term. The periods for adverse event tabulation will be from dose administration up to next dose administration if a further dose is given, and from dose administration to EOS for the last dose administration of a patient.
Determination of pharmacodynamic effect by means of biomarkers | Day 1 and Day 43
  Biomarker data from serum bone formation biomarkers: procollagen type I N-terminal propeptide, procollagen type I C-terminal propeptide, osteocalcin, and bone-specific alkaline phosphatase, and from serum bone resporption mbiomarkers: C-telopeptides of type I collagen cross-links, and N-telopeptides of type I collagen cross-links will be reported as concentration results, measured using a specific assay with a working range defined by the Lower limit of quantification and Upper limit of quantification. It will be considered a sign for efficacy, if any of the above show significant (2-sided, alpha=0.05) increase versus baseline in the BPS804 group on day 43.
Change in Z-score from baseline to Day 141 | Day 1 and Day 141
  Bone mineral density will be assessed by dual-energy X-ray absorptiometry of the lumbar spine. Analysis will include four vertebral levels from L1 to L4. Individual vertebral levels may be excluded due to artifact. Bone mineral density Z-scores will be used as these are a comparison of a patient's BMD to that of a patient of the same age, sex, and ethnicity. The comparison of change from baseline with the matching change in the reference group will be done by 2-sample t-tests (1-sided). It will be considered a sign for efficacy, if any of the above show significant (2-sided, alpha=0.05) increase versus baseline in the BPS804 group on day 141.

SECONDARY OUTCOMES:
Determination of the serum concentration-time profiles of BPS804 | Day 1 (prior to administration and 3x after administration) and Days 2, 8, 15 (2x), 16, 29 (4x), 30, 36, 43, 57, 85, 113,141
  Individual and overlaying individual serum concentration-time profiles of BPS804 will be constructed from the serial sampling on Day 1 (prior to administration and 3x after administration) and Days 2, 8, 15 (2x), 16, 29 (4x), 30, 36, 43, 57, 85, 113,141. In addition arithmetic and geometric mean serum concentration-time profiles of BPS804 will be constructed from the above data points.
Determination of the area under the serum concentration-time curve from time zero to the end of the dosing interval tau after the first dose | Day 1 (prior to administration and 3x after administration) and Days 2, and 8
  The area under the serum concentration-time curve from time zero to the end of the dosing interval tau after the first dose will be derived using using non-compartmental methods from data collected on Day 1 (4x) and Days 2, and 8.
Determination of the maximal concentration after the first dose | Day 1 (prior to administration and 3x after administration) and Days 2, and 8
  The maximal concentration after the first dose will be derived using using non-compartmental methods from data collected Day 1 (4x) and Days 2, and 8.
Determination of the time of maximal concentration after the first dose | Day 1 (prior to administration and 3x after administration) and Days 2, and 8
  The time of maximal concentration after the first dose will be derived using using non-compartmental methods from data collected Day 1 (4x) and Days 2, and 8.
Determination of the maximal concentration after the second dose | Day 15 (prior to administration and 1x after administration) and Day 16
  The maximal concentration after the second dose will be derived using using non-compartmental methods from data collected from days 15 (2x) and 16.
Determination of the time of maximal concentration after the second dose | Day 15 (prior to administration and 1x after administration) and Day 16
  The time of maximal concentration after the second dose will be derived using using non-compartmental methods from data collected from days 15 (2x) and 16.
Determination of the area under the serum concentration-time curve from time zero to infinity after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The area under the serum concentration-time curve from time zero to the end of the dosing interval tau after the third dose will be derived using non-compartmental methods from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141.
Determination of the area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration after the third dose will be derived using non-compartmental methods from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141.
Determination of the area under the serum concentration-time curve from time zero to the end of the dosing interval tau after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The area under the serum concentration-time curve from time zero to the end of the dosing interval tau after the third dose will be derived using non-compartmental methods from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141.
Determination of the maximal serum concentration after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The maximal serum concentration after the third dose will be derived using using non-compartmental methods from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141.
Determination of the time of maximal concentration after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The time of maximal concentration after the third dose will be derived using using non-compartmental methods from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141.
Determination of the terminal elimination half-life after the third dose | Days 29 (prior to administration and 3x after administration) and 30, 36, 43, 57, 85, 113, and 141
  The terminal elimination half-life after the third dose will be derived from data collected on Days 29 (4x), 30, 36, 43, 57, 85, 113, and 141 using a compound-specific modeling approach.
Determination of the concentration of total sclerostin in serum | Screening, Days 1, 8, 15, 29, 36, 43, 57, 85, 113, 141
  The function of sclerostin is described as an endogenous negative regulator of bone formation. Total serum sclerostin will be measured from samples collected at screening and on days 1, 8, 15, 29, 36, 43, 57, 85, 113, and 141
Immunogenicity evaluation in serum | Days 1, 29, 85, and 141
  Immunogenicity will only be assessed in patients randomized to the treatment group. Anti-BPS804 antibodies will be measured in human serum on Days 1, 29, 85, and 141 An immunogenicity positive patient at end of study will be followed up until anti-BPS804 antibody levels are back to levels measured on Day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (6):
- United States (2):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Miramar, Florida
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Würzburg, Germany

REFERENCES:
- [Background] Glorieux FH. Osteogenesis imperfecta. Best Pract Res Clin Rheumatol. 2008 Mar;22(1):85-100. doi: 10.1016/j.berh.2007.12.012. PMID 18328983